CLINICAL TRIAL: NCT03696485
Title: A Prospective, Single Center, Open Label, Dose Escalation Phase I/IIa Study to Assess the Safety and Efficacy of an Intrathecal Administration of SCM-010 in Subjects With Secondary Progressive Multiple Sclerosis (SPMS)
Brief Title: Study to Assess the Safety and Efficacy of an IT Administration of SCM-010 in SPMS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to sponsor decision
Sponsor: Stem Cell Medicine Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPMS-SCM-010
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: Secondary Progressive Multiple Sclerosis (SPMS), safety
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: low dose (Experimental): One intrathecal (IT) administration of SCM-010 at baseline visit
  Interventions: Biological: SCM-010
- group 2: high dose (Experimental): One intrathecal (IT) administration of SCM-010 at baseline visit
  Interventions: Biological: SCM-010

INTERVENTIONS:
Biological: SCM-010 — SCM-010 is comprised of adipose derived expanded mesenchymal cells (ADSC), suspended in Plasma-Lyte and intended for intrathecal (IT) administration.

SUMMARY:
Prospective, single center, open label, phase I/IIa escalating dose study. To evaluate the safety and efficacy of escalating doses of SCM-010 in subjects with SPMS.

DETAILED DESCRIPTION:
Twelve (12) SPMS subjects will be enrolled in this study in two dose cohorts. Each subject will receive SCM- 010 by intrathecal (IT) administration at baseline and will be followed up for 24 weeks for efficacy and 48 weeks for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (18-60 years of age) diagnosed with SPMS.
2. SPMS defined as relapsing-remitting disease followed by progression of disability independent of or not explained by multiple sclerosis (MS) relapses for at least 2 years.
3. Subjects should be ambulatory with an EDSS score of 3-6.5 (inclusive) at screening and baseline visits.
4. Subjects should be able to go through a lipoaspiration procedure, evaluated by the study's plastic surgeon.
5. Women capable of child bearing must have a negative urine pregnancy test at screening and baseline visits.
6. Subjects must use an adequate contraceptive method throughout the study.
7. Coagulation tests including INR, PTT and prothrombin time (PT) within normal range.
8. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
9. Ability to provide written informed consent.

Exclusion Criteria:

1. Relapsing remitting multiple sclerosis (RRMS) or primary progressive multiple sclerosis (PPMS) as defined by the revised McDonald criteria.
2. Any chronic central nervous system (CNS) disease other than SPMS.
3. Clinical relapse within 3 months prior to study entry.
4. Subjects diagnosed with any systemic autoimmune disease.
5. Contraindications or inability to undergo lumbar puncture (LP) procedure and or intrathecal administration.
6. Severe anemia (hemoglobin < 10 g/dL).
7. Abnormal renal function (serum creatinine more than 1.5xULN or creatinine clearance <30 ml/min).
8. Tested positive for HIV, hepatitis (HBV and HCV).
9. Known as positive for VDRL and/or tuberculosis.
10. Active malignant disease of any kind. However, a patient, who has had a malignant disease in the past, was treated and is currently disease - free for at least 7 years, may be considered eligible. In this case the sponsor medical expert approval is required.
11. Previous cell therapy treatment.
12. Previous total body irradiation or total lymphoid irradiation.
13. Previous use of natalizumab or any anti-B cell agent within 6 months prior to screening.
14. Previous use of immunosuppressant including Mitoxantrone, Alemtuzumab, Cladribine or any other cytotoxic agent.
15. Previous use of Fingolimod or Dimethyl Fumarate within 2 months prior to screening. Subjects who were treated with any of these medications will be excluded if they do not have a lymphocyte count within normal range at screening.
16. Previous use of Teriflunomide within 12 months if no accelerated elimination procedure was used.
17. Previous treatment with immunomodulators (including IFNβ 1a and 1b, and IV Immunoglobulin (IVIG) or Glatiramer Acetate (GA) within 2 months prior to screening.
18. A known history of hypersensitivity to one of following: Vancomycin, Cephalosporin, Cephamycin or beta-lactam antibacterial agent (penicillins, monobactams, carbapenems).
19. A known history of sensitivity to Gadolinium.
20. Inability to successfully undergo MRI scanning.
21. Treatment with any kind of steroids or ACTH during the last 30 days prior to screening.
22. Subjects with clotting disorders or receiving treatment with anticoagulants.
23. Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Principle Investigator, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
24. Subjects with BMI < 20.
25. Pregnant or breast-feeding women.
26. Known or suspected drug or alcohol abuse.
27. Participation in any investigational drug study within 6 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) reported during the trial | 48 weeks
  Safety data will be collected following the one IT administration of SCM-010 at baseline visit

SECONDARY OUTCOMES:
Change in MRI scans from baseline | 24 weeks
  Changes in lesions from baseline MRI scan.
Change from baseline in EDSS score | 24 weeks
  The Expanded Disability Status Scale (EDSS) will be measured during the study. range of the scale 0-10
Time to Confirmed Disease Progression (CDP) | 24 weeks
  CDP for an individual subject is defined as at least 3-months confirmed EDSS increase from baseline.
  The Expanded Disability Status Scale (EDSS) will be measured during the study. range of the scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Karni, Dr., Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel